CLINICAL TRIAL: NCT03004404
Title: A Partially Randomised, Single-blind, Placebo-controlled Trial to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Doses of BI 730357 Administered as Oral Solution and Tablets to Healthy Subjects, and a Randomized, Open-label, Single-dose, Three-way Cross-over Bioavailability Comparison of BI 730357 as Tablet Versus Oral Solution and Tablet With and Without Food
Brief Title: To Assess Safety, Tolerability and Pharmacokinetics of BI 730357 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1407.1; 2016-003047-11 (EudraCT Number)
Record Dates: First submitted 2016-12-23; First posted 2016-12-28 (Estimated); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant

ARMS (16):
- SRD part-Dose group 1: BI 730357 PfOS 2 mg Fasted (Experimental): Participants were administered on Day 1 a single oral dose of 2 milligram (mg) of BI 730357 powder for reconstitution of an oral solution (PfoS) reconstituted in solvent for oral solution 2 milliliter (mL) (Macrogol 400 (Polyethylene glycol 400) together with about 240 milliliter (mL) of water in fasted state.
  One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 730357
- Placebo (Placebo Comparator): This arm comprises all placebo treated participants in trial part SRD, regardless of the dose group in which they were treated. Participants of the first cohort of each dose group (DG) were not randomized. In the second cohort of each DG participants were assigned to active treatment or placebo in a 3:1 allocation ratio.
  Interventions: Drug: Placebo
- SRD part-Dose group 2: BI 730357 PfOS 8 mg Fasted (Experimental): Participants were administered on Day 1 a single oral dose of 8 milligram (mg) of BI 730357 powder for reconstitution of an oral solution (PfoS) reconstituted in solvent for oral solution 8 milliliter (mL) (Macrogol 400 (Polyethylene glycol 400) together with about 240 milliliter (mL) of water in fasted state.
  One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 730357
- SRD part-Dose group 3: BI 730357 tablet 25 mg Fasted (Experimental): Participants were administered on Day 1 a single oral dose of 25 milligram (mg) of BI 730357 film-coated tablet together with about 240 milliliter (mL) of water in fasted state. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 730357
- SRD part-Dose group 4: BI 730357 tablet 50 mg Fasted (Experimental): Participants were administered on Day 1 a single oral dose of 50 milligram (mg) of BI 730357 film-coated tablet together with about 240 milliliter (mL) of water in fasted state. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 730357
- SRD part-Dose group 5: BI 730357 tablet(s) 100 mg Fasted (Experimental): Participants were administered on Day 1 a single oral dose of 100 milligram (mg) of BI 730357 film-coated tablets (2x50mg) together with about 240 milliliter (mL) of water in fasted state. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 730357
- SRD part-Dose group 6: BI 730357 tablet(s) 200 mg Fasted (Experimental): Participants were administered on Day 1 a single oral dose of 200 milligram (mg) of BI 730357 film-coated tablets (4x50mg) together with about 240 milliliter (mL) of water in fasted state. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 730357
- SRD part-Dose group 7: BI 730357 tablet(s) 400 mg Fasted (Experimental): Participants were administered on Day 1 a single oral dose of 200 milligram (mg) of BI 730357 film-coated tablets (8x50mg) together with about 240 milliliter (mL) of water in fasted state. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 730357
- SRD part-Dose group 8-9: BI 730357 tablet(s) 400 mg Fed (Experimental): The same participants conformed the Dose group (DG) 8 and DG 9. DG 8: Participants were administered on Day 1 a single oral dose of 200 milligram (mg) of BI 730357 film-coated tablets (8x50mg) together with about 240 milliliter (mL) of water, 30 minutes (min) prior dose administration the participants consumed a standard continental breakfast.
  DG 9: Participants were administered on Day 1 a single oral dose of 200 milligram (mg) of BI 730357 film-coated tablets (8x50mg) together with about 240 milliliter (mL) of water, 30 minutes (min) prior dose administration the participants consumed a standard high fat breakfast.
  Both treatment periods were separated by a wash-out phase of at least 14 days between drug administration of DG 8 and DG 9. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 730357
- SRD part-Dose group 10: BI 730357 tablet(s) 800 mg Fed (Experimental): Participants were administered on Day 1 a single oral dose of 200 milligram (mg) of BI 730357 film-coated tablets (16x50mg) together with about 240 milliliter (mL) of water, 30 minutes (min) prior dose administration the participants consumed a standard high fat breakfast. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 730357
- BA Part: R/T2/T1 (Experimental): Participants were orally administered 25 mg of BI 730357 as film-coated tablet (Reference treatment R) in fasted state.
  Followed by 25 mg of BI 730357 film-coated tablet in a fed state (test treatment T2), a high-fat, high-calorie breakfast was served 30 min before dose administration.
  Participants received 25 mg of BI 730357 powder for reconstitution of an oral solution (PfOS) reconstituted in solvent for oral solution 2.5 milliliter (mL) (Macrogol 400 (Polyethylene glycol 400) (test treatment T1) in fasted state.
  The 3 treatments were administered with 240 mL of water and were separated by a washout period of at least 8 days. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 730357
- BA Part: R/T1/T2 (Experimental): Participants were orally administered 25 mg of BI 730357 as film-coated tablet (Reference treatment R) in fasted state.
  Participants received 25 mg of BI 730357 powder for reconstitution of an oral solution (PfOS) reconstituted in solvent for oral solution 2.5 milliliter (mL) (Macrogol 400 (Polyethylene glycol 400) (test treatment T1) in fasted state.
  Followed by 25 mg of BI 730357 film-coated tablet in a fed state (test treatment T2), a high-fat, high-calorie breakfast was served 30 min before dose administration.
  The 3 treatments were administered with 240 mL of water and were separated by a washout period of at least 8 days. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 730357
- BA Part: T2/R/T1 (Experimental): Participants were orally administered 25 mg of BI 730357 film-coated tablet in a fed state (test treatment T2), a high-fat, high-calorie breakfast was served 30 min before dose administration.
  Followed by 25 mg of BI 730357 as film-coated tablet (Reference treatment R) in fasted state.
  Participants received 25 mg of BI 730357 powder for reconstitution of an oral solution (PfOS) reconstituted in solvent for oral solution 2.5 milliliter (mL) (Macrogol 400 (Polyethylene glycol 400) (test treatment T1) in fasted state.
  The 3 treatments were administered with 240 mL of water and were separated by a washout period of at least 8 days. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 730357
- BA Part: T2/T1/R (Experimental): Participants were orally administered 25 mg of BI 730357 film-coated tablet in a fed state (test treatment T2), a high-fat, high-calorie breakfast was served 30 min before dose administration.
  Participants received 25 mg of BI 730357 powder for reconstitution of an oral solution (PfOS) reconstituted in solvent for oral solution 2.5 milliliter (mL) (Macrogol 400 (Polyethylene glycol 400) (test treatment T1) in fasted state.
  Followed by 25 mg of BI 730357 as film-coated tablet (Reference treatment R) in fasted state.
  The 3 treatments were administered with 240 mL of water and were separated by a washout period of at least 8 days. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 730357
- BA Part: T1/R/T2 (Experimental): Participants received 25 mg of BI 730357 powder for reconstitution of an oral solution (PfOS) reconstituted in solvent for oral solution 2.5 milliliter (mL) (Macrogol 400 (Polyethylene glycol 400) (test treatment T1) in fasted state.
  Followed by 25 mg of BI 730357 as film-coated tablet (Reference treatment R) in fasted state.
  Participants were orally administered 25 mg of BI 730357 film-coated tablet in a fed state (test treatment T2), a high-fat, high-calorie breakfast was served 30 min before dose administration.
  The 3 treatments were administered with 240 mL of water and were separated by a washout period of at least 8 days. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 730357
- BA Part: T1/T2/R (Experimental): BA Part: T1/T2/R Participants received 25 mg of BI 730357 powder for reconstitution of an oral solution (PfOS) reconstituted in solvent for oral solution 2.5 milliliter (mL) (Macrogol 400 (Polyethylene glycol 400) (test treatment T1) in fasted state.
  Participants were orally administered 25 mg of BI 730357 film-coated tablet in a fed state (test treatment T2), a high-fat, high-calorie breakfast was served 30 min before dose administration.
  Followed by 25 mg of BI 730357 as film-coated tablet (Reference treatment R) in fasted state.
  The 3 treatments were administered with 240 mL of water and were separated by a washout period of at least 8 days. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 730357

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: BI 730357 — powder for reconstitution of an oral solution (PfoS)
  Arms: BA Part: R/T1/T2; BA Part: R/T2/T1; BA Part: T1/R/T2; BA Part: T1/T2/R; BA Part: T2/R/T1; BA Part: T2/T1/R; SRD part-Dose group 1: BI 730357 PfOS 2 mg Fasted; SRD part-Dose group 2: BI 730357 PfOS 8 mg Fasted
Drug: BI 730357 — BI 730357 film-coated tablet
  Arms: BA Part: R/T1/T2; BA Part: R/T2/T1; BA Part: T1/R/T2; BA Part: T1/T2/R; BA Part: T2/R/T1; BA Part: T2/T1/R; SRD part-Dose group 10: BI 730357 tablet(s) 800 mg Fed; SRD part-Dose group 3: BI 730357 tablet 25 mg Fasted; SRD part-Dose group 4: BI 730357 tablet 50 mg Fasted; SRD part-Dose group 5: BI 730357 tablet(s) 100 mg Fasted; SRD part-Dose group 6: BI 730357 tablet(s) 200 mg Fasted; SRD part-Dose group 7: BI 730357 tablet(s) 400 mg Fasted; SRD part-Dose group 8-9: BI 730357 tablet(s) 400 mg Fed

SUMMARY:
The primary objective of the Single Rising Dose (SRD) part (trial part 1) is to investigate the safety and tolerability of BI 730357 in healthy subjects following oral administration of single rising doses after fasting and/or non-fasting conditions. The secondary objective is the exploration of the pharmacokinetics (PK) including dose proportionality, and pharmacodynamics of BI 730357 after single dosing.

The objective of the Bioavailability (BA) part (trial part 2) will be to explore the relative bioavailability of tablet fasted versus oral solution fasted and the influence of food on the bioavailability of tablet fasted versus tablet fed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male according to the Investigator's assessment, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (incl.)
* Body Mass index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the Investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the Investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the Investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc (corrected QT) interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the Investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

In addition, the following trial-specific exclusion criteria apply:

- Male subjects with Women of childbearing potential (WOCBP) partner who are unwilling to use male contraception (condom or sexual abstinence) from the first administration of trial medication until 30 days after last administration of trial medication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had two parts, single rising dose (SRD): partially randomized, single-blind, placebo-controlled, parallel group design to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of BI 730357. Bioavailability/food effect (BA/FE) part: Single dose, randomised, open-label, intra-individual three-way crossover to investigate the relative BA of the tablet formulation versus oral solution as well as the influence of food on the bioavailability of the tablet formulation.
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were not to be randomised to trial drug if any of the specific entry criteria was violated.
Groups:
- Placebo: This arm comprises all placebo treated participants in trial part SRD, regardless of the dose group in which they were treated. Participants of the first cohort of each dose group (DG) were not randomized. In the second cohort of each DG participants were assigned to active treatment or placebo in a 3:1 allocation ratio.
  Participants were administered on Day 1 a single oral dose of matching placebo, for dose group (DG) 1-2 the matching placebo was solvent for oral solution containing Macrogol 400 (Polyethylene glycol 400) on a volume identical to dose group of active treatment, for DG 3-7 the matching placebo were single oral film-coated tablet(s) with about 240 milliliter (mL) of water on fasted state. For DG 8-10 the matching placebo were single oral film-coated tablet(s) with about 240 milliliter (mL) of water on fed state, 30 minutes (min) prior dose administration the participants consumed a standard high fat breakfast/continental breakfast depending on dose group. One authorized employee of the trial site was witness of the administration of the trial medication.
- BA Part: T1/T2/R: Participants received 25 mg of BI 730357 powder for reconstitution of an oral solution (PfOS) reconstituted in solvent for oral solution 2.5 milliliter (mL) (Macrogol 400 (Polyethylene glycol 400) (test treatment T1) in fasted state.
  Participants were orally administered 25 mg of BI 730357 film-coated tablet in a fed state (test treatment T2), a high-fat, high-calorie breakfast was served 30 min before dose administration.
  Followed by 25 mg of BI 730357 as film-coated tablet (Reference treatment R) in fasted state.
  The 3 treatments were administered with 240 mL of water and were separated by a washout period of at least 8 days. One authorized employee of the trial site was witness of the administration of the trial medication.
Period: Period 1
Arm/Group | Placebo | SRD Part-Dose Group 1: BI 730357 PfOS 2 mg Fasted | SRD Part-Dose Group 2: BI 730357 PfOS 8 mg Fasted | SRD Part-Dose Group 3: BI 730357 Tablet 25 mg Fasted | SRD Part-Dose Group 4: BI 730357 Tablet 50 mg Fasted | SRD Part-Dose Group 5: BI 730357 Tablet(s) 100 mg Fasted | SRD Part-Dose Group 6: BI 730357 Tablet(s) 200 mg Fasted | SRD Part-Dose Group 7: BI 730357 Tablet(s) 400 mg Fasted | SRD Part-Dose Group 8-9: BI 730357 Tablet(s) 400 mg Fed | SRD Part-Dose Group 10: BI 730357 Tablet(s) 800 mg Fed | BA Part: R/T2/T1 | BA Part: R/T1/T2 | BA Part: T2/R/T1 | BA Part: T2/T1/R | BA Part: T1/R/T2 | BA Part: T1/T2/R
Started | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Placebo | SRD Part-Dose Group 1: BI 730357 PfOS 2 mg Fasted | SRD Part-Dose Group 2: BI 730357 PfOS 8 mg Fasted | SRD Part-Dose Group 3: BI 730357 Tablet 25 mg Fasted | SRD Part-Dose Group 4: BI 730357 Tablet 50 mg Fasted | SRD Part-Dose Group 5: BI 730357 Tablet(s) 100 mg Fasted | SRD Part-Dose Group 6: BI 730357 Tablet(s) 200 mg Fasted | SRD Part-Dose Group 7: BI 730357 Tablet(s) 400 mg Fasted | SRD Part-Dose Group 8-9: BI 730357 Tablet(s) 400 mg Fed | SRD Part-Dose Group 10: BI 730357 Tablet(s) 800 mg Fed | BA Part: R/T2/T1 | BA Part: R/T1/T2 | BA Part: T2/R/T1 | BA Part: T2/T1/R | BA Part: T1/R/T2 | BA Part: T1/T2/R
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 2 | 2 | 2 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 3
Arm/Group | Placebo | SRD Part-Dose Group 1: BI 730357 PfOS 2 mg Fasted | SRD Part-Dose Group 2: BI 730357 PfOS 8 mg Fasted | SRD Part-Dose Group 3: BI 730357 Tablet 25 mg Fasted | SRD Part-Dose Group 4: BI 730357 Tablet 50 mg Fasted | SRD Part-Dose Group 5: BI 730357 Tablet(s) 100 mg Fasted | SRD Part-Dose Group 6: BI 730357 Tablet(s) 200 mg Fasted | SRD Part-Dose Group 7: BI 730357 Tablet(s) 400 mg Fasted | SRD Part-Dose Group 8-9: BI 730357 Tablet(s) 400 mg Fed | SRD Part-Dose Group 10: BI 730357 Tablet(s) 800 mg Fed | BA Part: R/T2/T1 | BA Part: R/T1/T2 | BA Part: T2/R/T1 | BA Part: T2/T1/R | BA Part: T1/R/T2 | BA Part: T1/T2/R
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The Treated set (TS) included all subjects from the Randomised set (RS) who were documented to have taken at least 1 dose of trial medication. The TS for the SRD part included 72 subjects. The TS for the BA part included all 12 treated subjects.
Groups:
- BA Part: In the BA part of the trial, subjects were randomised to 6 treatment sequences. All subjects were administered BI 730357 as tablet in fasted condition (R), as oral solution in fasted condition (T1), and as tablet after a standardised high-fat breakfast (T2). The 3 treatments were separated by a wash-out period of at least 8 days between trial drug administrations. One authorized employee of the trial site was witness of the administration of the trial medication.
- Total: Total of all reporting groups
Arm/Group | Placebo | SRD Part-Dose Group 1: BI 730357 PfOS 2 mg Fasted | SRD Part-Dose Group 2: BI 730357 PfOS 8 mg Fasted | SRD Part-Dose Group 3: BI 730357 Tablet 25 mg Fasted | SRD Part-Dose Group 4: BI 730357 Tablet 50 mg Fasted | SRD Part-Dose Group 5: BI 730357 Tablet(s) 100 mg Fasted | SRD Part-Dose Group 6: BI 730357 Tablet(s) 200 mg Fasted | SRD Part-Dose Group 7: BI 730357 Tablet(s) 400 mg Fasted | SRD Part-Dose Group 8-9: BI 730357 Tablet(s) 400 mg Fed | SRD Part-Dose Group 10: BI 730357 Tablet(s) 800 mg Fed | BA Part | Total
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 84
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Treated set
  Years | 32.3 (6.3) | 36.8 (4.5) | 33.0 (6.5) | 30.7 (6.7) | 30.2 (8.7) | 31.3 (5.0) | 30.2 (7.9) | 34.5 (5.9) | 30.8 (7.0) | 31.7 (5.5) | 35.3 (8.6) | 32.6 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Treated Set
  Participants
    Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Male | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — TS
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 84
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Treated Set
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    White | 17 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 83
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug-related Adverse Events (AEs)
Description: Percentage of subjects with adverse reactions, assessed by investigator-defined drug-related adverse events (AEs) are reported.
  Fed1 means intake of continental breakfast; fed2 means intake of high-fat breakfast. The 400 mg tablet fed1 and fed2 treatments were administered to the same participants.
Time Frame: SRD 1-7, 10: From first drug administration until end of trial (EOT), up to 13 days. SRD 8-9: From first drug administration until end of trial (EOT), up to 27 days. BA: From first drug administration until end of trial (EOT), up to 41 days.
Population: Treated set (TS): This subject set included all subjects from the Randomised set (RS) who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Measure: Number; unit: Percentage of participants
Groups:
- SRD Part-Dose Group 8: BI 730357 Tablets(s) 400 mg Fed1: Participants were administered on Day 1 a single oral dose of 200 milligram (mg) of BI 730357 film-coated tablets (8x50mg) together with about 240 milliliter (mL) of water, 30 minutes (min) prior dose administration the participants consumed a standard continental breakfast. One authorized employee of the trial site was witness of the administration of the trial medication.
- SRD Part-Dose Group 9: BI 730357 Tablets(s) 400 mg Fed2: Participants were administered on Day 1 of period 2 a single oral dose of 200 milligram (mg) of BI 730357 film-coated tablets (8x50mg) together with about 240 milliliter (mL) of water, 30 minutes (min) prior dose administration the participants consumed a standard high fat breakfast. One authorized employee of the trial site was witness of the administration of the trial medication.
- BA Part: BI 730357 Tablet 25 mg Fasted (R): Participants were orally administered 25 mg of BI 730357 as film-coated tablet (Reference treatment R) together with about 240 mL of water in fasted state. One authorized employee of the trial site was witness of the administration of the trial medication.
- BA Part: BI 730357 PfOS 25 mg Fasted (T1): Participants received 25 mg of BI 730357 powder for reconstitution of an oral solution (PfOS) reconstituted in solvent for oral solution 2.5 milliliter (mL) (Macrogol 400 (Polyethylene glycol 400) (test treatment T1) together with about 240 mL of water in fasted state. One authorized employee of the trial site was witness of the administration of the trial medication.
- BA Part: BI 730357 Tablet 25 mg Fed (T2): Participants were orally administered 25 mg of BI 730357 film-coated tablet in a fed state (test treatment T2) together with about 240 mL of water, a high-fat, high-calorie breakfast was served 30 min before dose administration. One authorized employee of the trial site was witness of the administration of the trial medication.
Arm/Group | Placebo | SRD Part-Dose Group 1: BI 730357 PfOS 2 mg Fasted | SRD Part-Dose Group 2: BI 730357 PfOS 8 mg Fasted | SRD Part-Dose Group 3: BI 730357 Tablet 25 mg Fasted | SRD Part-Dose Group 4: BI 730357 Tablet 50 mg Fasted | SRD Part-Dose Group 5: BI 730357 Tablet(s) 100 mg Fasted | SRD Part-Dose Group 6: BI 730357 Tablet(s) 200 mg Fasted | SRD Part-Dose Group 7: BI 730357 Tablet(s) 400 mg Fasted | SRD Part-Dose Group 8: BI 730357 Tablets(s) 400 mg Fed1 | SRD Part-Dose Group 9: BI 730357 Tablets(s) 400 mg Fed2 | SRD Part-Dose Group 10: BI 730357 Tablet(s) 800 mg Fed | BA Part: BI 730357 Tablet 25 mg Fasted (R) | BA Part: BI 730357 PfOS 25 mg Fasted (T1) | BA Part: BI 730357 Tablet 25 mg Fed (T2)
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 11 | 12 | 12
Percentage of participants | 5.6 | 0.0 | 16.7 | 0.0 | 0.0 | 16.7 | 16.7 | 0.0 | 0.0 | 20.0 | 0.0 | 0.0 | 0.0 | 0.0

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 730357 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-inf)
Description: Area under the concentration-time curve of BI 730357 in plasma over the time interval from 0 extrapolated to infinity is reported.
  Fed1 means intake of continental breakfast; fed2 means intake of high-fat breakfast. The 400 mg tablet fed1 and fed2 treatments were administered to the same subjects.
Time Frame: SRD & BA Part: Within 3 hours (h) prior administration, and 0.5h, 1.0h, 1.5h, 2.0h, 2.5h, 3.0h, 4.0h, 5.0h, 6.0h, 8.0h, 10.0h, 12.0h, 24.0h, 34.0h, 48.0h, 72.0h, 96.0h and 168.0h after drug administration
Population: Pharmacokinetic set (PKS): The PKS included all subjects who were treated with BI 730357 and who provided at least 1 secondary PK endpoint (AUC0-∞ or Cmax) that was not excluded due to a protocol violation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol*hour/liter (nmol*h/L)
Groups:
- SRD Part-Dose Group 9: BI 730357 Tablets(s) 400 mg Fed2: Participants were administered on Day 1 a single oral dose of 200 milligram (mg) of BI 730357 film-coated tablets (8x50mg) together with about 240 milliliter (mL) of water, 30 minutes (min) prior dose administration the participants consumed a standard high fat breakfast. One authorized employee of the trial site was witness of the administration of the trial medication.
Arm/Group | SRD Part-Dose Group 1: BI 730357 PfOS 2 mg Fasted | SRD Part-Dose Group 2: BI 730357 PfOS 8 mg Fasted | SRD Part-Dose Group 3: BI 730357 Tablet 25 mg Fasted | SRD Part-Dose Group 4: BI 730357 Tablet 50 mg Fasted | SRD Part-Dose Group 5: BI 730357 Tablet(s) 100 mg Fasted | SRD Part-Dose Group 6: BI 730357 Tablet(s) 200 mg Fasted | SRD Part-Dose Group 7: BI 730357 Tablet(s) 400 mg Fasted | SRD Part-Dose Group 8: BI 730357 Tablets(s) 400 mg Fed1 | SRD Part-Dose Group 9: BI 730357 Tablets(s) 400 mg Fed2 | SRD Part-Dose Group 10: BI 730357 Tablet(s) 800 mg Fed | BA Part: BI 730357 Tablet 25 mg Fasted (R) | BA Part: BI 730357 PfOS 25 mg Fasted (T1) | BA Part: BI 730357 Tablet 25 mg Fed (T2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 11 | 12 | 12
nanomol*hour/liter (nmol*h/L) | 399.0 (35.0) | 1550.0 (27.8) | 3730.0 (36.4) | 6990.0 (52.7) | 10700.0 (60.2) | 18300.0 (28.0) | 30800.0 (36.8) | 44800.0 (41.5) | 50700.0 (57.5) | 77900.0 (38.3) | 4240.0 (45.0) | 5390.0 (43.8) | 5370.0 (44.6)
Statistical Analysis 1: Comparison: SRD Part-Dose Group 3: BI 730357 Tablet 25 mg Fasted vs SRD Part-Dose Group 4: BI 730357 Tablet 50 mg Fasted vs SRD Part-Dose Group 5: BI 730357 Tablet(s) 100 mg Fasted vs SRD Part-Dose Group 6: BI 730357 Tablet(s) 200 mg Fasted vs SRD Part-Dose Group 7: BI 730357 Tablet(s) 400 mg Fasted; In the SRD part of the trial, dose proportionality for AUC0-inf was assessed in the 25 mg to 400 mg dose groups (BI 730357 tablets administered under fasted conditions) using a power model (regression model applied to log-transformed data); Test type: Other; Slope = 0.7480, 95% CI 2-sided [0.5959 to 0.9001], Standard Error of Mean 0.0743 — Standard error of the mean is actually standard error of the slope. Based on the estimate for the slope parameter, a two sided 95% confidence interval for the slope was computed. Perfect dose proportionality would correspond to a slope of 1
Statistical Analysis 2: Comparison: SRD Part-Dose Group 8: BI 730357 Tablets(s) 400 mg Fed1 vs SRD Part-Dose Group 9: BI 730357 Tablets(s) 400 mg Fed2; Relative bioavailability of AUC0-inf for the SRD part was performed to test the effect of food intake on the PK of 400 mg BI 730357 tablets. The intra-individual comparison of fed conditions was done using an Analysis of Variance (ANOVA) model on the logarithmic scale; Test type: Other; Ratio T/R = 118.71, 90% CI 2-sided [94.57 to 149.03], Standard Error of Mean 1.11 — Standard error of the mean is the geometric standard error of the mean. The geometric mean ratio was calculated as: tablet 400mg fed1 (T)/400mg fed2(R), T/R
Statistical Analysis 3: Comparison: BA Part: BI 730357 Tablet 25 mg Fasted (R) vs BA Part: BI 730357 PfOS 25 mg Fasted (T1); Estimation of relative bioavailability of AUC0-inf was based on ANOVA model on the logarithmic scale, included effects: 'sequence', 'period' and 'treatment' as fixed and 'subjects within sequences' as random; Test type: Other; Geometric mean ratio T1/R (%) = 124.79, 90% CI 2-sided [116.858 to 133.255], Standard Error of Mean 1.036 — Standard error of the mean is actually geometric standard error of the mean. The geometric mean ratio was calculated as: oral solution in fasted state (test treatment T1)/tablet in fasted state (reference treatment R), T1/R; Relative bioavailability of BI 730357 for Oral solution (PfOS) fasted (T1) vs. tablet fasted (R) was assessed by the point estimators (geometric means) of the intra-subject ratio of Auc0-inf and their two-sided 90% confidence intervals . No hypothesis was tested
Statistical Analysis 4: Comparison: BA Part: BI 730357 Tablet 25 mg Fasted (R) vs BA Part: BI 730357 Tablet 25 mg Fed (T2); [analysis description as in outcome 2, analysis 3]; Test type: Other; Geometric mean ratio T2/R (%) = 125.17, 90% CI 2-sided [112.89 to 138.80], Standard Error of Mean 1.06 — Standard error of the mean is actually geometric standard error of the mean. The geometric mean ratio was calculated as: tablet in fed state (test treatment T2)/tablet in fasted state (reference treatment R), T2/R; Relative bioavailability of BI 730357 for tablet fed (T2) vs. tablet fasted (R) was assessed by the point estimators (geometric means) of the intra-subject ratio of AUC0-inf and their two-sided 90% confidence intervals . No hypothesis was tested

3. Secondary Outcome: Maximum Measured Concentration of BI 730357 in Plasma (Cmax)
Description: Maximum measured concentration of BI 730357 in plasma is reported.
  Fed1 means intake of continental breakfast; Fed2 means intake of high-fat breakfast. The 400 mg tablet fed1 and fed2 treatments were administered to the same subjects.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol / liter (nmol/L)
Arm/Group | SRD Part-Dose Group 1: BI 730357 PfOS 2 mg Fasted | SRD Part-Dose Group 2: BI 730357 PfOS 8 mg Fasted | SRD Part-Dose Group 3: BI 730357 Tablet 25 mg Fasted | SRD Part-Dose Group 4: BI 730357 Tablet 50 mg Fasted | SRD Part-Dose Group 5: BI 730357 Tablet(s) 100 mg Fasted | SRD Part-Dose Group 6: BI 730357 Tablet(s) 200 mg Fasted | SRD Part-Dose Group 7: BI 730357 Tablet(s) 400 mg Fasted | SRD Part-Dose Group 8: BI 730357 Tablets(s) 400 mg Fed1 | SRD Part-Dose Group 9: BI 730357 Tablets(s) 400 mg Fed2 | SRD Part-Dose Group 10: BI 730357 Tablet(s) 800 mg Fed | BA Part: BI 730357 Tablet 25 mg Fasted (R) | BA Part: BI 730357 PfOS 25 mg Fasted (T1) | BA Part: BI 730357 Tablet 25 mg Fed (T2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 11 | 12 | 12
nanomol / liter (nmol/L) | 32.9 (39.4) | 154.0 (28.9) | 103.0 (31.7) | 173.0 (41.9) | 284.0 (30.7) | 433.0 (27.6) | 755.0 (37.4) | 1270.0 (17.5) | 1900.0 (30.2) | 2470.0 (15.7) | 133.0 (31.4) | 380.0 (27.4) | 235.0 (28.5)
Statistical Analysis 1: Comparison: SRD Part-Dose Group 3: BI 730357 Tablet 25 mg Fasted vs SRD Part-Dose Group 4: BI 730357 Tablet 50 mg Fasted vs SRD Part-Dose Group 5: BI 730357 Tablet(s) 100 mg Fasted vs SRD Part-Dose Group 6: BI 730357 Tablet(s) 200 mg Fasted vs SRD Part-Dose Group 7: BI 730357 Tablet(s) 400 mg Fasted; In the SRD part of the trial, dose proportionality for Cmax was assessed in the 25 mg to 400 mg dose groups (BI 730357 tablets administered under fasted conditions) using a power model (regression model applied to log-transformed data); Test type: Other; Slope = 0.7065, 95% CI 2-sided [0.5863 to 0.8267], Standard Error of Mean 0.0587 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: SRD Part-Dose Group 8: BI 730357 Tablets(s) 400 mg Fed1 vs SRD Part-Dose Group 9: BI 730357 Tablets(s) 400 mg Fed2; Relative bioavailability of the Cmax for the SRD part was performed to test the effect of food intake on the PK of 400 mg BI 730357 tablets. The intra-individual comparison of fed conditions was done using an ANOVA model on the logarithmic scale; Test type: Other; Ratio T/R = 151.22, 90% CI 2-sided [122.781 to 186.248], Standard Error of Mean 1.107 — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: BA Part: BI 730357 Tablet 25 mg Fasted (R) vs BA Part: BI 730357 PfOS 25 mg Fasted (T1); Estimation of relative bioavailability of Cmax based on ANOVA model on the logarithmic scale, included effects: 'sequence', 'period' and 'treatment' as fixed and 'subjects within sequences' as random; Test type: Other; Geometric mean ratio T1/R (%) = 293.21, 90% CI 2-sided [259.044 to 331.891], Standard Error of Mean 1.069 — Standard error of the mean is the geometric standard error of the mean. The geometric mean ratio was calculated as: oral solution in fasted state (test treatment T1)/tablet in fasted state (reference treatment R), T1/R; Relative bioavailability of BI 730357 for Oral solution (PfOS) fasted (T1) vs. tablet fasted (R) was assessed by the point estimators (geometric means) of the intra-subject ratio of Cmax and their two-sided 90% confidence intervals . No hypothesis was tested
Statistical Analysis 4: Comparison: BA Part: BI 730357 Tablet 25 mg Fasted (R) vs BA Part: BI 730357 Tablet 25 mg Fed (T2); Estimation of relative bioavailability of Cmax was based on ANOVA model on the logarithmic scale, included effects: 'sequence', 'period' and 'treatment' as fixed and 'subjects within sequences' as random; Test type: Other; Geometric mean ratio T2/R (%) = 180.53, 90% CI 2-sided [162.369 to 200.732], Standard Error of Mean 1.059 — Standard error of the mean is the geometric standard error of the mean. The geometric mean ratio was calculated as: tablet in fed state (test treatment T2)/tablet in fasted state (reference treatment R), T2/R; Relative bioavailability of BI 730357 for tablet fasted (T2) vs. tablet fasted (R) was assessed by the point estimators (geometric means) of the intra-subject ratio of Cmax and their two-sided 90% confidence intervals . No hypothesis was tested

ADVERSE EVENTS:
Time Frame: SRD 1-7, 9-10: From first drug administration until end of trial (EOT), up to 13 days. SRD 8: From first drug administration until end of trial (EOT), up to 14 days. BA per treatment: From first drug administration until end of trial (EOT), up to 14 days.
Description: Treated set (TS): This subject set included all subjects from the Randomised set (RS) who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Arm/Group | Placebo | SRD Part-Dose Group 1: BI 730357 PfOS 2 mg Fasted | SRD Part-Dose Group 2: BI 730357 PfOS 8 mg Fasted | SRD Part-Dose Group 3: BI 730357 Tablet 25 mg Fasted | SRD Part-Dose Group 4: BI 730357 Tablet 50 mg Fasted | SRD Part-Dose Group 5: BI 730357 Tablet(s) 100 mg Fasted | SRD Part-Dose Group 6: BI 730357 Tablet(s) 200 mg Fasted | SRD Part-Dose Group 7: BI 730357 Tablet(s) 400 mg Fasted | SRD Part-Dose Group 8: BI 730357 Tablets(s) 400 mg Fed1 | SRD Part-Dose Group 9: BI 730357 Tablets(s) 400 mg Fed2 | SRD Part-Dose Group 10: BI 730357 Tablet(s) 800 mg Fed | BA Part: BI 730357 Tablet 25 mg Fasted (R) | BA Part: BI 730357 PfOS 25 mg Fasted (T1) | BA Part: BI 730357 Tablet 25 mg Fed (T2)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/11 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/11 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/18 | 3/6 | 3/6 | 1/6 | 2/6 | 4/6 | 2/6 | 3/6 | 5/6 | 3/5 | 1/6 | 2/11 | 2/12 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | SRD Part-Dose Group 1: BI 730357 PfOS 2 mg Fasted (N=6) | SRD Part-Dose Group 2: BI 730357 PfOS 8 mg Fasted (N=6) | SRD Part-Dose Group 3: BI 730357 Tablet 25 mg Fasted (N=6) | SRD Part-Dose Group 4: BI 730357 Tablet 50 mg Fasted (N=6) | SRD Part-Dose Group 5: BI 730357 Tablet(s) 100 mg Fasted (N=6) | SRD Part-Dose Group 6: BI 730357 Tablet(s) 200 mg Fasted (N=6) | SRD Part-Dose Group 7: BI 730357 Tablet(s) 400 mg Fasted (N=6) | SRD Part-Dose Group 8: BI 730357 Tablets(s) 400 mg Fed1 (N=6) | SRD Part-Dose Group 9: BI 730357 Tablets(s) 400 mg Fed2 (N=5) | SRD Part-Dose Group 10: BI 730357 Tablet(s) 800 mg Fed (N=6) | BA Part: BI 730357 Tablet 25 mg Fasted (R) (N=11) | BA Part: BI 730357 PfOS 25 mg Fasted (T1) (N=12) | BA Part: BI 730357 Tablet 25 mg Fed (T2) (N=12)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medical device site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device failure (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT03004404/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/04/NCT03004404/SAP_001.pdf